CLINICAL TRIAL: NCT05443594
Title: A Prospective Single Arm Open Label Study of the FARAPULSE Pulsed Field Ablation System in Subjects With Persistent Atrial Fibrillation
Acronym: ADVANTAGE AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 92836802
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pulsed Field Ablation (Phase 1) (Experimental): PHASE 1 only
  Interventions: Device: Phase 1: FARAPULSE Ablation System
- Pulsed Field Ablation (Phase 2) (Experimental): PHASE 2 only
  Interventions: Device: Phase 2: FARAPULSE Ablation System

INTERVENTIONS:
Device: Phase 1: FARAPULSE Ablation System — PHASE 1: Pulsed Field Ablation to isolate the Pulmonary Veins and Posterior Wall using the FARAPULSE Ablation System.
  Arms: Pulsed Field Ablation (Phase 1)
Device: Phase 2: FARAPULSE Ablation System — PHASE 2: Pulsed Field Ablation to isolate the Pulmonary Veins, Posterior Wall and Cavo-Tricuspid Isthmus using the FARAPULSE Ablation System.
  Arms: Pulsed Field Ablation (Phase 2)

SUMMARY:
The objective of the ADVANTAGE AF Study is to establish the safety and effectiveness of the FARAPULSE Pulsed Field Ablation System (FARAPULSE PFA System) for treatment of drug resistant, symptomatic persistent atrial fibrillation (PersAF).

ELIGIBILITY:
[PHASE 1] --------------------------------------------

Inclusion Criteria:

1. Age ≥ 18 years of age, or older if specified by local law
2. Subjects have symptomatic, documented, drug-resistant, Persistent AF, defined as:

   a. Documented: at a minimum a physician's note confirming the arrhythmia symptoms and durations AND, within 180 days of Enrollment Date, either: i. A 24-hour continuous ECG recording confirming continuous AF OR ii. Two ECGs from any regulatory cleared rhythm monitoring device showing continuous AF taken at least 7 days apart b. Drug-resistant: effectiveness failure of, intolerance to, or specific contraindication to at least one (1) AAD (Class I or III).

   c. Persistent: continuous AF for > 7 days and ≤ 365 days
3. Subjects who are willing and capable of providing informed consent
4. Subjects who are willing and capable of participating in all testing associated with this clinical investigation at an approved clinical investigational center

Exclusion Criteria:

1. Any of the following atrial conditions:

   1. Left atrial anteroposterior diameter ≥ 5.5 cm, or if LA diameter not available, non-indexed volume >100 ml (by MRI, CT or TTE report or physician note)
   2. Any prior atrial endocardial, epicardial or surgical ablation procedure for arrhythmia, other than right sided cavotricuspid isthmus ablation or for right sided SVT
   3. Current atrial myxoma
   4. Any PV abnormality, stenosis, or stenting (common and middle PVs are admissible)
   5. Current left atrial thrombus
2. Cardiovascular exclusions - Any of the following CV conditions:

   a. History of sustained ventricular tachycardia or any ventricular fibrillation b. AF that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes c. Current or anticipated pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices, interatrial baffle, closure device, patch, or patent foramen ovale occluder, LA appendage closure, device or occlusion, active implantable loop recorder or insertable cardiac monitor at the time of ablation d. Valvular disease that is any of the following: i. Symptomatic ii. Causing or exacerbating congestive heart failure iii. Associated with abnormal LV function or hemodynamic measurements e. Hypertrophic cardiomyopathy f. Any prosthetic heart valve, ring or repair including balloon aortic valvuloplasty g. Any IVC filter, known inability to obtain vascular access or other contraindication to femoral access h. Rheumatic heart disease i. Congenital heart disease with any clinically significant residual anatomic or conduction abnormality j. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months
3. Any of the following conditions at baseline (Section7.5):

   1. Heart failure associated with NYHA Class III or IV
   2. LVEF < 40%
   3. Uncontrolled hypertension (SBP > 160 mmHg or DBP > 95 mmHg on two (2) BP measurements at baseline assessment
4. Any of the following events within 90 days of the Consent Date:

   1. Myocardial infarction (MI), unstable angina or coronary intervention
   2. Any cardiac surgery
   3. Heart failure hospitalization
   4. Pericarditis or symptomatic pericardial effusion
   5. Gastrointestinal bleeding
   6. Stroke, TIA, or intracranial bleeding
   7. Any non-neurologic thromboembolic event
   8. Carotid stenting or endarterectomy
5. Thrombocytosis, thrombocytopenia, disorder of blood clotting or bleeding diathesis
6. Contraindication to, or unwillingness to use, systemic anticoagulation
7. Patients who have not been on anticoagulation therapy for at least 4 weeks prior to the ablation procedure
8. Women of childbearing potential who are pregnant, lactating, not using medical birth control or who are planning to become pregnant during the anticipated study period
9. Health conditions that in the investigator's medical opinion would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation, including but not limited to:

   1. Body Mass Index (BMI) > 42.0
   2. Solid organ or hematologic transplant, or currently being evaluated for a transplant
   3. Any prior history or current evidence of hemi-diaphragmatic paralysis or paresis.
   4. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or requiring supplemental oxygen
   5. Renal insufficiency if an estimated glomerular filtration rate (eGFR) is < 30 mL / min / 1.73 m2, or with any history of renal dialysis or renal transplant
   6. Active malignancy or history of treated malignancy within 24 months of enrollment (other than cutaneous basal cell or squamous cell carcinoma)
   7. Clinically significant gastrointestinal problems involving the esophagus or stomach including severe or erosive esophagitis, uncontrolled gastric reflux, gastroparesis, esophageal candidiasis or active gastroduodenal ulceration
   8. Active systemic infection
   9. COVID-19 disease

   i. Current confirmed, active COVID-19 disease ii. Current positive test for SARS-CoV-2 iii. Confirmed COVID-19 disease not clinically resolved at least 3 months prior to the Consent Date j. Uncontrolled diabetes mellitus or a recorded HgbA1c > 8.0% in the 90 days prior to the Consent Date k. Untreated diagnosed obstructive sleep apnea with apnea hypopnea index classification of severe (>30 pauses per hour)
10. Predicted life expectancy less than one (1) year
11. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the Sponsor to determine eligibility

[PHASE 2] --------------------------------------------

Inclusion Criteria:

1. Age ≥ 18 years of age, or older if specified by local law
2. Subjects have symptomatic, documented, drug-resistant, Persistent AF, defined as:

   a. Documented: at a minimum a physician's note confirming the arrhythmia symptoms and durations AND, within 180 days of Enrollment Date, either: i. A 24-hour continuous ECG recording confirming continuous AF OR ii. Two ECGs from any regulatory cleared rhythm monitoring device showing continuous AF taken at least 7 days apart b. Drug-resistant: effectiveness failure of, intolerance to, or specific contraindication to at least one (1) AAD (Class I or III).

   c. Persistent: continuous AF for > 7 days and ≤ 365 days
3. Subjects who are willing and capable of providing informed consent
4. Subjects who are willing and capable of participating in all testing associated with this clinical investigation at an approved clinical investigational center

Exclusion Criteria:

1. Any of the following atrial conditions:

   1. Left atrial anteroposterior diameter ≥ 5.5 cm, or if LA diameter not available, non-indexed volume >100 ml (by MRI, CT or TTE report or physician note)
   2. Any prior atrial endocardial, epicardial or surgical ablation procedure for arrhythmia, other than right sided cavotricuspid isthmus ablation or for right sided SVT
   3. Current atrial myxoma
   4. Any PV abnormality, stenosis, or stenting (common and middle PVs are admissible)
   5. Current left atrial thrombus
2. Cardiovascular exclusions - Any of the following CV conditions:

   1. History of sustained ventricular tachycardia or any ventricular fibrillation
   2. AF that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes
   3. Current or anticipated pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices, interatrial baffle, closure device, patch, or patent foramen ovale occluder, LA appendage closure, device or occlusion, active implantable loop recorder or insertable cardiac monitor at the time of ablation
   4. Valvular disease that is any of the following:

   i. Symptomatic ii. Causing or exacerbating congestive heart failure iii. Associated with abnormal LV function or hemodynamic measurements e. Hypertrophic cardiomyopathy f. Any prosthetic heart valve, ring or repair including balloon aortic valvuloplasty g. Any IVC filter, known inability to obtain vascular access or other contraindication to femoral access h. Rheumatic heart disease i. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months j. Nitroglycerin intolerance: Known adverse drug reaction to nitroglycerin k. Coronary disease: Known severe non-revascularizable coronary disease l. Stents: Pre-existing right coronary artery stent
3. Any of the following conditions at baseline (Section7.5):

   1. Heart failure associated with NYHA Class III or IV
   2. LVEF < 40%
   3. Uncontrolled hypertension (SBP > 160 mmHg or DBP > 95 mmHg on two (2) BP measurements at baseline assessment
   4. Ventricular dysfunction: Right ventricular dysfunction
4. Any of the following events within 90 days of the Consent Date:

   1. Myocardial infarction (MI), unstable angina or coronary intervention
   2. Any cardiac surgery
   3. Heart failure hospitalization
   4. Pericarditis or symptomatic pericardial effusion
   5. Gastrointestinal bleeding
   6. Stroke, TIA, or intracranial bleeding
   7. Any non-neurologic thromboembolic event
   8. Carotid stenting or endarterectomy
5. Thrombocytosis, thrombocytopenia, disorder of blood clotting or bleeding diathesis
6. Contraindication to, or unwillingness to use, systemic anticoagulation
7. Patients who have not been on anticoagulation therapy for at least 4 weeks prior to the ablation procedure
8. Women of childbearing potential who are pregnant, lactating, not using medical birth control or who are planning to become pregnant during the anticipated study period
9. Health conditions that in the investigator's medical opinion would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation, including but not limited to:

   1. Body Mass Index (BMI) > 42.0
   2. Solid organ or hematologic transplant, or currently being evaluated for a transplant
   3. Any prior history or current evidence of hemi-diaphragmatic paralysis or paresis.
   4. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or requiring supplemental oxygen
   5. Renal insufficiency if an estimated glomerular filtration rate (eGFR) is < 30 mL / min / 1.73 m2, or with any history of renal dialysis or renal transplant
   6. Active malignancy or history of treated malignancy within 24 months of enrollment (other than cutaneous basal cell or squamous cell carcinoma)
   7. Clinically significant gastrointestinal problems involving the esophagus or stomach including severe or erosive esophagitis, uncontrolled gastric reflux, gastroparesis, esophageal candidiasis or active gastroduodenal ulceration
   8. Active systemic infection
   9. COVID-19 disease

   i. Current confirmed, active COVID-19 disease ii. Current positive test for SARS-CoV-2 iii. Confirmed COVID-19 disease not clinically resolved at least 3 months prior to the Consent Date j. Uncontrolled diabetes mellitus or a recorded HgbA1c > 8.0% in the 90 days prior to the Consent Date k. Untreated diagnosed obstructive sleep apnea with apnea hypopnea index classification of severe (>30 pauses per hour) l. Medication Use: Required use of phosphodiesterase inhibitors within 24 hours of the ablation procedure
10. Predicted life expectancy less than one (1) year
11. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the Sponsor to determine eligibility
12. Any of the following congenital conditions:

    1. Congenital heart disease: Congenital heart disease with any clinically significant residual anatomic or conduction abnormality
    2. Methemoglobinemia: History of known congenital methemoglobinemia
    3. G6PD deficiency: History of known G6PD deficiency
13. Contraindication to ICM insertion: Patients who cannot tolerate a subcutaneous, chronically-inserted LUX-Dx device
14. LUX-Dx longevity: Patients with a LUX-Dx device inserted > 6 months prior to enrollment with an estimated longevity of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (44):
- United States (40):
  - Grandview Medical Center-Hospital, Birmingham, Alabama
  - Banner University Medical Center Phoenix-Hospital, Phoenix, Arizona
  - Arrhythmia Research Group-Research Facility, Jonesboro, Arkansas
  - Scripps Memorial Hospital-Hospital, La Jolla, California
  - Cedars - Sinai Medical Center-Hospital, Los Angeles, California
  - University of California, San Francisco-Hospital, San Francisco, California
  - Emory University Hospital-Hospital, Atlanta, Georgia
  - St. Lukes Idaho Cardiology Associates-Hospital, Boise, Idaho
  - Northwestern University-Hospital, Evanston, Illinois
  - St. John's Hospital-Hospital, Springfield, Illinois
  - St. Vincent's Hospital-Hospital, Indianapolis, Indiana
  - Mercy Hospital Medical Center-Hospital, West Des Moines, Iowa
  - University of Kansas Hospital-Hospital, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Johns Hopkins Hospital - East Baltimore Campus, Baltimore, Maryland
  - Massachusetts General Hospital-Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital-Hospital, Boston, Massachusetts
  - Lahey Clinic Hospital-Hospital, Burlington, Massachusetts
  - St. Luke's Hospital of Kansas City-Hospital, Kansas City, Missouri
  - Catholic Medical Center-Hospital, Manchester, New Hampshire
  - Valley Hospital-Hospital, Ridgewood, New Jersey
  - NYU Langone Health Heart Rhythm Center, New York, New York
  - Weill Cornell Medical University-Hospital, New York, New York
  - Mount Sinai Medical Center-Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital-Hospital, Roslyn, New York
  - Bethesda North Hospital-Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation-Hospital, Cleveland, Ohio
  - OhioHealth Research and Innovation Institute - Riverside Methodist Hospital-Hospital, Columbus, Ohio
  - Doylestown Hospital-Hospital, Doylestown, Pennsylvania
  - UPMC Heart and Vascular Institute Harrisburg, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania-Hospital, Philadelphia, Pennsylvania
  - Trident Medical Center-Hospital, Charleston, South Carolina
  - St. Thomas Research Institute, LLC-Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center-Hospital, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research-Hospital, Austin, Texas
  - Orion Medical - Gulf Commerce Drive, Houston, Texas
  - Christus Trinity Mother Frances Health System-Hospital, Tyler, Texas
  - Sentara Norfolk General Hospital-Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Health System-Hospital, Richmond, Virginia
- UZ Brussel (AZ VUB)-Hospital, Brussels, Belgium
- Canada (2):
  - McGill University Health Centre-Hospital, Montreal, Quebec
  - Institut universitaire de Cardiologie et de Pneumologie de Quebec-Hospital, Ste-Foy, Quebec
- Clinica Universidad de Navarra-Hospital, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerstenfeld EP, Schmidt B, Natale A, Nair D, Saliba W, Verma A, Sommer P, Metzner A, Dewland TA, Moss JD, Amin A, Champagne J, Cuoco F, Hounshell T, Issa Z, Turagam M, Brose R, Schwartz T, Raybuck JD, Garlitski A, Mansour M, Reddy VY. Pulsed Field Ablation vs Standard Radiofrequency Ablation for Typical Atrial Flutter: ADVANTAGE AF Trial Substudy. J Am Coll Cardiol. 2026 Feb 6:S0735-1097(26)00055-0. doi: 10.1016/j.jacc.2025.12.081. Online ahead of print. PMID 41653174
- [Derived] Matsumoto K, van Bragt KA, Kueffer FJ, Mburu W, Tarakji KG. Indirect treatment comparison of two pulsed field ablation systems for the treatment of persistent atrial fibrillation. J Interv Card Electrophysiol. 2025 Sep 10. doi: 10.1007/s10840-025-02124-6. Online ahead of print. PMID 40928625
- [Derived] Reddy VY, Gerstenfeld EP, Schmidt B, Nair D, Natale A, Saliba W, Verma A, Sommer P, Metzner A, Turagam M, Weiner S, Champagne J, Garcio-Bolao I, Calkins H, Olson J, Issa Z, Winner M, Su W, Tomassoni G, Kim J, Hook B, Delurgio DB, Gibson DN, Daccarett M, Patel C, Bhalla K, Shehata M, Harding JD, Cheung JW, Raybuck JD, Roelke S, Schwartz T, Sutton BS, Mansour M; ADVANTAGE-AF Investigators. Pulsed Field Ablation for Persistent Atrial Fibrillation: 1-Year Results of ADVANTAGE AF. J Am Coll Cardiol. 2025 May 6;85(17):1664-1678. doi: 10.1016/j.jacc.2025.03.515. PMID 40306839
- [Derived] Reddy VY, Gerstenfeld EP, Schmidt B, Andrade JG, Nair D, Natale A, Saliba W, Sommer P, Metzner A, Verma A, Hounshell T, Amin A, Gentlesk P, Weiner S, Cuoco FA, Kim J, Turagam MK, Tomassoni G, Patel C, Issa Z, Shehata M, Anderson AM, Stoltz TJ, Raybuck JD, Schwartz T, Sutton BS, Mansour M; ADVANTAGE AF Investigators. Pulsed Field Ablation of Persistent Atrial Fibrillation With Continuous Electrocardiographic Monitoring Follow-Up: ADVANTAGE AF Phase 2. Circulation. 2025 Jul 8;152(1):27-40. doi: 10.1161/CIRCULATIONAHA.125.074485. Epub 2025 Apr 24. PMID 40273320

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulsed Field Ablation (Phase 1): PHASE 1 only
  Phase 1: FARAPULSE Ablation System - Pulsed Field Ablation (PFA) to isolate the Pulmonary Veins and Posterior Wall using the FARAWAVE PFA Catheter.
- Pulse Field Ablation (Phase 2): Phase 2 only
  Phase 2: FARAPULSE Ablation System - Pulsed Field Ablation (PFA) to isolate the Pulmonary Veins and Posterior Wall using the FARAWAVE PFA Catheter and FARAPOINT PFA Catheter for cavo-tricuspid isthmus (CTI) ablation.
Period: Overall Study
Arm/Group | Pulsed Field Ablation (Phase 1) | Pulse Field Ablation (Phase 2)
Started | 355 | 314
Completed | 325 | 290
Not Completed | 30 | 24

BASELINE CHARACTERISTICS:
Population: This patient population are the 260 Non-Roll in subjects in Phase 1 and 255 subjects in Phase 2 who received treatment with the PFA System.
Groups:
- Pulsed Field Ablation (Phase 1) Non-Roll In Treatment Subjects: PHASE 1 only
  Phase 1: FARAPULSE Ablation System - Pulsed Field Ablation (PFA) to isolate the Pulmonary Veins and Posterior Wall using the FARAWAVE PFA Catheter.
- Pulsed Field Ablation (Phase 2) Non-Roll In Treatment Subjects: Phase 2 only
  Phase 2: FARAPULSE Ablation System - Pulsed Field Ablation (PFA) to isolate the Pulmonary Veins and Posterior Wall using the FARAWAVE PFA Catheter and FARAPOINT PFA Catheter for cavo-tricuspid isthmus (CTI) ablation.
- Total: Total of all reporting groups
Arm/Group | Pulsed Field Ablation (Phase 1) Non-Roll In Treatment Subjects | Pulsed Field Ablation (Phase 2) Non-Roll In Treatment Subjects | Total
Number analyzed (Participants) | 260 | 255 | 515
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (9.3) | 66.7 (9.3) | 66.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 73 | 153
  Male | 180 | 182 | 362
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 211 | 245 | 456
  Unknown or Not Reported | 45 | 5 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 209 | 241 | 450
  Other | 0 | 1 | 1
  Unknown or Not Report | 45 | 5 | 50
Height (cm) [Mean (Standard Deviation); unit: cm] | 175.8 (9.7) | 177.6 (10.6) | 176.7 (10.2)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 94.3 (19.7) | 98 (20.3) | 96.1 (20.1)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (5.3) | 30.9 (5.3) | 30.7 (5.3)
Resting Heart Rate (bpm) [Mean (Standard Deviation); unit: bpm] | 74 (18.3) | 76.8 (18.7) | 75.4 (18.5)
Systolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 129.9 (16.6) | 129.8 (16.6) | 129.8 (16.6)
Diastolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 77.5 (10.0) | 77.6 (10.3) | 77.5 (10.1)
Left Ventricular Ejection Fraction (%) [Mean (Standard Deviation); unit: % blood ejected from the left ventricle] | 57.2 (6.9) | 56.6 (6.7) | 56.9 (6.8)
LA Diameter (cm) [Mean (Standard Deviation); unit: cm] | 4.3 (0.6) | 4.3 (0.6) | 4.3 (0.6)
LA Volume (mL) [Mean (Standard Deviation); unit: mL] | 65.1 (24.6) | 65.5 (19.3) | 65.2 (23.0)
NYHA [Number; unit: participants] — New York Heart Association (NYHA) Heart Failure Classification based on the severity of heart failure symptoms as assessed by the clinician - progressively ranging from no heart failure to Class IV heart failure.
  participants
    No Heart Failure | 173 | 140 | 313
    Class I | 42 | 52 | 94
    Class II | 44 | 63 | 107
    Class III | 0 | 0 | 0
    Class IV | 0 | 0 | 0
CHA₂DS₂-VASc Score [Count of Participants; unit: Participants] — The CHA2DS2-VASc Score for Atrial Fibrillation Stroke Risk - is a point-based system that considers several risk factors, and the total score helps determine the likelihood of stroke (i.e., the stroke risk for patients with atrial fibrillation). The higher the score the higher the risk.
  Participants
    1 | 47 | 46 | 93
    2 | 59 | 68 | 127
    3 | 64 | 65 | 129
    4 | 43 | 37 | 80
    5 | 12 | 16 | 28
    6 | 4 | 1 | 5
    7 | 0 | 1 | 1
    0 | 31 | 21 | 52

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint (PSE): Event Rate of Safety Events Post Procedure
Description: Phase 1:
  Through 7 Days:
  * Myocardial infarction
  * Stroke
  * Transient Ischemic Attack (TIA)
  * Peripheral or organ thromboembolism
  * Pulmonary edema
  * Unresolved phrenic nerve palsy / paresis
  * Vascular access complications
  * Heart block
  * Gastric motility / pyloric spasm disorders
  Through 30 Days:
  * Cardiac tamponade / perforation
  * Pericarditis
  Through 360 Days Post-Procedure:
  * PV stenosis
  * Atrio-esophageal fistula
  Phase 2
  Through 7 Days:
  * Myocardial infarction
  * Stroke
  * Transient Ischemic Attack (TIA)
  * Peripheral or organ thromboembolism
  * Pulmonary edema
  * Unresolved phrenic nerve palsy / paresis
  * Vascular access complications
  * Heart block
  * Gastric motility / pyloric spasm disorders
  Through 30 Days:
  * Death
  * Cardiac tamponade / perforation
  * Pericarditis
  * Any PFA system related PFA procedure-related cardiovascular or pulmonary adverse event
  Through 90 Days:
  * PV stenosis
  * Atrio-esophageal fistula
Time Frame: Phase 1 Index Procedure through 360 Days | Phase 2 Index Procedure through 90 Days (per protocol Primary Safety Endpoint requirements)
Population: Adverse Events reported for subjects were reviewed and adjudicated for meeting Safety Endpoint criteria by an independent physician Clinical Events Committee.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | Pulsed Field Ablation (Phase 1) Non-Roll In Treatment Subjects | Pulsed Field Ablation (Phase 2) Non-Roll In Treatment Subjects
Number analyzed (Participants) | 260 | 255
Percentage of participants | 2.3 [NA to 5.1] — One sided confidence interval | 2.4 [NA to 5.2] — One sided confidence interval

2. Primary Outcome: Primary Effectiveness Endpoint: Treatment Success Rate Through Day 360
Description: Includes both Acute Procedural Success and Chronic Success through Day 360.
Time Frame: Post-Blanking Period: Day 90 through Day 360
Population: Note: Phase 1 includes all Non-Roll in Treatment subjects. Phase 2 includes Non-Roll in Treatment subjects who received an Insertable Cardiac Monitor for arrhythmia recurrence monitoring.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Groups:
- Pulse Field Ablation (Phase 2) Non-Roll In Treatment Subject: Phase 2 only
  Phase 2: FARAPULSE Ablation System - Pulsed Field Ablation (PFA) to isolate the Pulmonary Veins and Posterior Wall using the FARAWAVE PFA Catheter and FARAPOINT PFA Catheter for cavo-tricuspid isthmus (CTI) ablation.
Arm/Group | Pulsed Field Ablation (Phase 1) Non-Roll In Treatment Subjects | Pulse Field Ablation (Phase 2) Non-Roll In Treatment Subject
Number analyzed (Participants) | 260 | 253
Percentage of participants | 63.5 [57.3 to NA] — One-sided confidence interval | 73.4 [67.5 to NA] — One-sided confidence interval

3. Other Pre Specified Outcome: Rate of Persistent AF Chronic Success
Description: Defined as the freedom from any of the following through the Day 360 Assessment after the Blanking Period, excluding documented CTI-dependent AFL for phase 1 and for Phase 2 excluding documented CTI-dependent AFL if the participant did not have a CTI ablation with a FARAPOINT PFA Catheter:
  1. Arrhythmia: Occurrence of any Detectable AF, AFL or AT
  2. Re-ablation: Any re-ablation for AF, AFL or AT
  3. Cardioversion: Any electrical cardioversion for AF, AFL or AT
  4. AAD Use: Use of a Non-Failed Class I / III AAD or amiodarone
Time Frame: Post-Blanking Period: Day 90 through Day 360
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pulsed Field Ablation (Phase 1) Non-Roll In Treatment Subjects | Pulsed Field Ablation (Phase 2) Non-Roll In Treatment Subjects
Number analyzed (Participants) | 260 | 253
Percentage of participants | 64.2 [58.1 to 70.1] | 73.4 [67.5 to 78.4]

4. Other Pre Specified Outcome: Rate of Persistent AF Acute Procedural Success
Description: * The isolation of all attempted PVs as clinically assessed at the end of the procedure by entrance block performed with or without adenosine testing, AND
  * The isolation of the left atrial PW as clinically assessed at the end of the procedure, performed with or without adenosine testing, via interrogation by multipolar diagnostic catheter or 3D electroanatomical mapping.
  * Use of an ablation catheter other than the FARAWAVE Pulse Field Ablation Catheter (i.e., use of a non-study catheter) to achieve Pulmonary Vein Isolation and Posterior Wall Isolation.
Time Frame: Assessed through Index Ablation Procedure
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pulsed Field Ablation (Phase 1) Non-Roll In Treatment Subjects | Pulsed Field Ablation (Phase 2) Non-Roll In Treatment Subjects
Number analyzed (Participants) | 260 | 253
Percentage of participants | 99.6 [97.9 to 100] | 99.6 [97.8 to 100]

5. Post Hoc Outcome: Freedom From Documented Symptomatic Recurrence and Intervention
Description: Freedom from symptomatic recurrence and intervention is Chronic Treatment Success, as defined for the Primary Effectiveness Endpoint, but excluding failure due to asymptomatic detectable AF, AFL, or AT.
Time Frame: Post-Blanking Period: Day 90 through Day 360
Population: Note: Freedom from Documented Symptomatic Recurrence and Intervention was a post-hoc analysis for the Phase 1 cohort and a pre-specified analysis for the Phase 2 cohort.
  Note: Phase 1 includes all Non-Roll in Treatment subjects. Phase 2 includes Non-Roll in Treatment subjects who received an Insertable Cardiac Monitor for arrhythmia recurrence monitoring.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | Pulsed Field Ablation (Phase 1) Non-Roll In Treatment Subjects | Pulsed Field Ablation (Phase 2) Non-Roll In Treatment Subjects
Number analyzed (Participants) | 260 | 253
Percentage of participants | 85.3 [80.3 to NA] — One sided confidence interval | 81.0 [75.5 to 85.3]

ADVERSE EVENTS:
Time Frame: Through Day 360
Arm/Group | Pulsed Field Ablation (Phase 1) Non-Roll In Treatment Subjects | Pulsed Field Ablation (Phase 2) Non-Roll In Treatment Subjects
All-Cause Mortality (participants affected / at risk) | 0/260 | 2/255
Serious Adverse Events (participants affected / at risk) | 44/260 | 53/255
Other Adverse Events (participants affected / at risk) | 82/260 | 76/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulsed Field Ablation (Phase 1) Non-Roll In Treatment Subjects (N=260) | Pulsed Field Ablation (Phase 2) Non-Roll In Treatment Subjects (N=255)
2nd degree AV block (Cardiac disorders) | 1 (1) | 0 (0)
Abnormal laboratory values (Surgical and medical procedures) | 3 (3) | 0 (0)
Adverse reaction-Medication (Surgical and medical procedures) | 1 (1) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 9 (10) | 10 (11)
Atrial Flutter (Cardiac disorders) | 1 (1) | 3 (3)
Atrial tachycardia/ Other SVT (AVRT, AVNRT, EAT) (Cardiac disorders) | 2 (2) | 1 (1)
Cancer (Infections and infestations) | 1 (1) | 1 (1)
Cerebrovascular Accident (CVA) (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular Accident (CVA)- Hemorrhagic (Nervous system disorders) | 1 (1) | 2 (2)
Coronary artery Disease (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery injury/ spasm (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea (Cardiac disorders) | 1 (1) | 0 (0)
Exacerbation of existing condition (General disorders) | 2 (2) | 0 (0)
Fluid volume overload (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 4 (5)
Genitourinary (Renal and urinary disorders) | 3 (4) | 2 (2)
Hematoma - Unrelated procedure/device (Vascular disorders) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 1 (1) | 0 (0)
Physical Trauma (General disorders) | 1 (1) | 1 (1)
Pleural effusion - unrelated procedure/ device (General disorders) | 1 (1) | 1 (1)
Post procedure infection/ sepsis (Infections and infestations) | 1 (1) | 1 (1)
Procedure related Anesthesia/ sedation (Surgical and medical procedures) | 1 (1) | 1 (1)
Procedure related Genitourinary/ renal (Surgical and medical procedures) | 4 (4) | 0 (0)
Procedure related heart failure (Surgical and medical procedures) | 3 (3) | 0 (0)
Procedure related hypotension (Surgical and medical procedures) | 1 (1) | 1 (1)
Procedure related Neurological (Non-TIA, non-stroke, dysphagia, speech disturbance/ dysarthria) (Surgical and medical procedures) | 1 (1) | 0 (0)
Procedure related Pulmonary (including cough, hemoptysis) (Surgical and medical procedures) | 2 (2) | 1 (1)
Psychological (Psychiatric disorders) | 1 (1) | 0 (0)
ST segment elevation (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 0 (0)
Thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Valvular damage/ valvular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
AV block (Transient) (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - Other (General disorders) | 0 (0) | 2 (2)
Dyspnea - Heart Failure (Cardiac disorders) | 0 (0) | 2 (2)
Embolism - Air (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head, Eyes, Ears, Nose, Throat (HEENT) (General disorders) | 0 (0) | 1 (2)
Hemolysis (laboratory confirmed) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hemolysis high suspicion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Hypertension/Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension/Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Impaired Mobility (Cardiac disorders) | 0 (0) | 1 (1)
Infection - Unrelated procedure/device (Infections and infestations) | 0 (0) | 2 (2)
Major bleeding/Hemorrhage requiring transfusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Myocardial infarction (Vascular disorders) | 0 (0) | 1 (1)
Myocardial perforation with tamponade (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neurological (Nervous system disorders) | 0 (0) | 1 (1)
Pericardial effusion - Unrelated procedure/device (Cardiac disorders) | 0 (0) | 1 (1)
Post-surgical pocket hemorrhage/bleeding/drainage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedure related Abnormal labs (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedure related Fatigue/Weakness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedure related Genitourinary (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedure related Renal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 5 (5)
Stroke (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vasovagal reaction (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulsed Field Ablation (Phase 1) Non-Roll In Treatment Subjects (N=260) | Pulsed Field Ablation (Phase 2) Non-Roll In Treatment Subjects (N=255)
Edema (General disorders) | 2 (2) | 0 (0)
AV block (permanent) (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 11 (13) | 8 (8)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia/ Other SVT(AVRT, AVNRT, EAT) (Cardiac disorders) | 3 (3) | 0 (0)
Chest pain - Ischemic (Vascular disorders) | 0 (0) | 1 (1)
Fatigue/ weakness (General disorders) | 1 (1) | 0 (0)
Hypertension/ hypertensive crisis (Cardiac disorders) | 2 (2) | 1 (1)
Multiple heart failure symptoms (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral edema - Heart Failure (General disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 6 (6)
Syncope (Cardiac disorders) | 1 (1) | 0 (0)
Cancer (General disorders) | 1 (1) | 1 (1)
Genitourinary (Renal and urinary disorders) | 3 (3) | 0 (0)
Localized infection (Infections and infestations) | 1 (1) | 0 (0)
Physical trauma (General disorders) | 1 (1) | 1 (1)
Psychological (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
1st degree AV block (Cardiac disorders) | 0 (0) | 2 (2)
Adverse reaction - Medication (General disorders) | 0 (0) | 2 (2)
Angina/Chest pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Atrial flutter, not specified (Cardiac disorders) | 3 (3) | 1 (1)
Bruising access site (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Cerebrovascular Accident (CVA) - Hemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Chest pain - Ischemic (General disorders) | 2 (2) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (1)
Edema (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Erosion (Product Issues) | 0 (0) | 1 (1)
Fever and/or virus (Infections and infestations) | 0 (0) | 1 (1)
Fluid volume overload (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 3 (3)
Headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heart Failure symptoms - Unspecified (Cardiac disorders) | 0 (0) | 3 (3)
Hematological (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Hemolysis (Laboratory confirmed) (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Hiccups (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Inadequate healing of incision site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Non-Sustained Ventricular Tachycardia (NSVT) (Cardiac disorders) | 0 (0) | 1 (1)
Non-symptomatic pericardial effusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Oozing/Bleeding (Injury, poisoning and procedural complications) | 7 (7) | 10 (10)
Pain (Non-cardiovascular) (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Pain cardiovascular (Non-ischemic) (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Phrenic nerve injury temporary (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pleural effusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedure infection/sepsis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedure wound discomfort (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Post -surgical infection (<=30 days post implant) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-surgical pocket hemorrhage/bleeding/drainage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedure related Abnormal labs (Injury, poisoning and procedural complications) | 2 (3) | 4 (4)
Procedure related Allergic reactions/Adverse drug reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedure related Anesthesia/Sedation (Injury, poisoning and procedural complications) | 11 (14) | 2 (2)
Procedure related Gastrointestinal (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Procedure related Genitourinary (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedure related Genitourinary/Renal (Injury, poisoning and procedural complications) | 13 (13) | 0 (0)
Procedure related Heart Failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedure related Hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedure related Hypotension (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Procedure related Neurological (Non-TIA, non-stroke, dysphagia, speech disturbance/dysarthria) (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Procedure related Pulmonary (including cough, hemoptysis) (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pulmonary edema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Symptomatic pericardial effusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vasovagal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Visual blurring/disturbances, Migraine (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT05443594/Prot_SAP_001.pdf